CLINICAL TRIAL: NCT02411240
Title: Air Pollution Reduction in the Elderly and Cardiovascular and Cognitive Outcomes, an Intervention Study
Brief Title: Air Pollution Reduction in the Elderly and Cardiovascular and Cognitive Outcomes
Acronym: ELIFA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Tim Nawrot, Associate professor, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ELIFA_TN
Record Dates: First submitted 2014-07-21; First posted 2015-04-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Beneficial Health Effects of Living in Filtered Air
Keywords: Air filtration; cardiovascular health; cognition; particulate matter; mitochondrial DNA
MeSH Terms: interventions — Air Filters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Air filtering in the living room (Other): GENANO tubes, GENANO Benelux; Heusen-Zolder, Belgium
  Interventions: Device: Air filtering

INTERVENTIONS:
Device: Air filtering — The air filter will be placed in the living room of the elderly people. The efficiency of this device has been tested and a drop of ultrafine particles of more then 70 % is achieved.
  Other Names: GENANO tubes, GENANO Benelux; Heusen-Zolder, Belgium

SUMMARY:
Short-term and chronic exposure to ambient levels of particulate matter (PM) is associated with increased morbidity and mortality related to respiratory and cardiovascular disease. Proposed biological pathways imply that particle-induced inflammation plays a role in activating the vascular endothelium and altering vascular function. Accumulating evidence suggests that outdoor air pollution has a significant impact on central nervous system health and disease and living in conditions with elevated air pollution has been linked to decreased cognitive function.

Only recently was shown that reductions in ambient levels of PM2.5 were associated with improvements in life expectancy. However, studies of the beneficial effects of improved indoor air quality on healthy humans are lacking.

With this project the investigators intend to study the effects of rooms with clean air in the elderly with the emphasis on cardiovascular and cognitive function. The investigators hypothesise that by means of air cleaning, controlled and reduced exposure has a positive effect on cardiovascular parameters such as blood pressure, heart rate variability, macro- and microcirculation and on neurobehavioral function. The investigators substantiate these outcomes with potential mechanisms of action at the transcript and epigenetic level as with hematological parameters, markers of inflammation, lipid and protein oxidation products and mitochondrial DNA damage. To achieve these goals there is a specific need to study the elderly, as they appear to have elevated susceptibility and have the largest attributable risk related to indoor PM, as they spend more time indoors. Suited concepts for study location are elderly homes ("service flats") and retirement homes.

The "ELiFA"-cohort stands for Elderly Living in Filtered Air consisting of an intervention study during 2-week periods of a pre-purification (baseline), active purification and a post purification period.

DETAILED DESCRIPTION:
1. Study Population and Design

   Persons living in ''service flats'' or retirement homes are healthy elderly who respectively live semi-independently or dependently. The elderly homes will be located in Flanders, Belgium. Persons are included if they are 65 years or older, not bedridden, non- smoker and able to give informed consent. This selection is made on the basis of the mental state of candidate participants, this primary selection is based on the advice of the directors or head nurses of the elderly homes.

   A documented minimental state examination (MMSE) will be performed and the participation of the candidates will depend on a priori determined criteria (score 23) and the ability of the possible participant to perform the NES tests (cognitive test), done a priori of enrolment. The project design is an intervention study of in total 6 weeks, starting with a baseline pre-purification period, a 2-week active purification period and a 2-week post purification period. Each participant is his/her own control, excluding confounding by factors that are stable within an individual over time but vary between participants.

   The device (GENANO tubes, GENANO Benelux; Heusen-Zolder, België) is placed in the living room of each apartment during the study period. These kinds of air purification devices are used in medical settings (cleanrooms, medical practice) and give us the opportunity to create a well-controlled experimental real life setting.

   Ultra fine particle (UFP) (Aerasense, Philips), PM10-2.5 and total suspended particulates (TSP) (Aerocet, MetOne) are monitored. Blood and urine are sampled every week in the morning at the same hour per participant to avoid problems due to diurnal variation. The participants will be asked to fill in a questionnaire. For the duration of the study, the investigators ask the participants to keep their windows closed.
2. Primary Endpoints The primary endpoints focus on changes in the cardiovascular en neurobiological function.

   2.1 Cardiovascular function. The cardiovascular measurements are conducted non-invasively and are wide ranging in order to comprehensively study these effects.

   2.1.1. Microvasculature: After pupillary dilation, digital images of both the retinas are obtained using a digital retinal camera (Canon CR-2 Digital Retinal Camera).

   2.1.2. Macro vasculature: The distensibility and intermedia thickness of the carotid artery are measured by echo-graphical imaging with the esaote MY LAB ™ ONE mobil device.

   2.1.3.Heart rate variability: With a mobile ECG sensor (Biopatch, Zephyr) the heart rate variability (HRV) is continuously monitored for several 24h periods during the 3 phases of the study.

   2.1.4. Blood pressure: Using Stabil-O-Graph devices the blood pressure is determined 5 consecutive times for every time point.

   2.2 Cognitive function The investigators assess the neurobehavioral function with the Neurobehavioral Evaluation System (NES-3). Neurobehavioral Evaluation System (NES) is a computerised battery of tests developed to study the neurological effects of an exposure to environmental agents. The investigators use the digit span test, the continuous performance and the Stroop test.
3. Secondary Endpoints The investigators delineate these outcomes with secondary endpoints to find potential mechanisms of action at the transcript and epigenetic level as with on haematological parameters, markers of inflammation and lipid and protein oxidation products and mitochondrial DNA damage.

3.1. Transcriptomics and Epigenetics The investigators study underlying mechanisms either by full transcriptome analysis and gene specific transcription patterns as well as by specific hypothesis driven microRNA studies. Epigenetic profiles are studied by gene specific methylation sequencing.

3.2. Haematological measurements, markers of inflammation, and oxidative stress.

The investigators measure hemoglobin, red blood cells, fibrinogen, platelets, coagulation factors (II + VII + X), IL-6 and urinary 8-oxo-7,8-dihydro-2'-deoxyguanosine (8-oxo-dG).

3.3. Mitochondrial DNA damage The investigators measure the mitochondrial DNA content relative to nuclear DNA by means of qPCR, which is a measure of DNA damage and can give an indication of the need to repair mitochondrial DNA damage. As this parameter is an early sensor of DNA-damage these samples will be collected from the whole blood tubes.

ELIGIBILITY:
Inclusion Criteria:

* The selection is made on the basis of the mental state of candidate participants, this primary selection is based on the advice of the directors or head nurses of the elderly homes, as in the investigators' previous studies (Jacobs et al., 2012).
* A documented minimental state examination (MMSE) will be performed and the participation of the candidates will depend on a priori determined criteria (score of 23) and the ability of the possible participant to perform the NES tests (cognitive test), done a priori of enrolment.

Exclusion Criteria:

* 65 years or older
* Non- smoker
* Not bed-ridden
* Able to give informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive endpoints as assessed by the Neurobehavioral Evaluation System (NES-3) | The cognitive outcome is performed weekly during the 6 week period, changes from baseline measurement are studied
  The investigators assess the neurobehavioral function with the Neurobehavioral Evaluation System (NES-3) (Baker et al., 1985, Kiciński et al., 2012). Neurobehavioral Evaluation System (NES) is a computerized battery of tests developed to study the neurological effects of an exposure to environmental agents. They use the digit span test, the continuous performance and the Stroop test.
Cardiovascular endpoint: Microvasculature | The cardiovascular outcome is performed weekly during the 6 week period, changes from baseline measurement are studied
  Microvasculature imaging is performed to establish changes in cardiovascular status due to living in filtered air. Microvasculature is measured by taking a digital picture of the retina vasculature using a digital retinal camera (Canon CR-2 Digital Retinal Camera), the diameter of the retinal vasculature is determined.
Cardiovascular endpoint: Macro vasculature (carotid intima media thickness) | The cardiovascular outcome is performed weekly during the 6 week period, changes from baseline measurement are studied
  Macro vasculature is determined to establish changes in cardiovascular status due to living in filtered air. Macro vasculature is determined by measuring the carotid intima media thickness using the esaote MY LAB ™ ONE mobil device.
Cardiovascular endpoint: Heart rate variability (24h) | The cardiovascular outcome is performed weekly during the 6 week period, changes from baseline measurement are studied
  Heart rate variability (hrv) measurements are performed to establish changes in cardiovascular status due to living in filtered air. Hrv (24h) is measured using a Zephyr biopatch attached to the chest.
Cardiovascular endpoint: Blood pressure | The cardiovascular outcome is performed weekly during the 6 week period, changes from baseline measurement are studied
  Blood pressure is measured to establish changes in cardiovascular status due to living in filtered air. Using Stabil-O-Graph devices the blood pressure is determined 5 consecutive times for every time point.

SECONDARY OUTCOMES:
Underlying mechanisms at the molecular level: Transcriptomics and Epigenetics | Weekly during the 6 week period, changes from baseline measurement are studied
  Underlying mechanisms are studied either by full transcriptome analysis and gene specific transcription patterns as well as by specific hypothesis driven microRNA studies. Epigenetic profiles are studied by gene specific methylation sequencing. This is a composite outcome studying the processes influencing gene-expression.
Underlying mechanisms at the molecular level: Markers of inflammation, and oxidative stress and haematological markers | Weekly during the 6 week period, changes from baseline measurement are studied
  The investigators measure hemoglobin, red blood cells, fibrinogen, platelets, coagulation factors (II + VII + X), IL-6 and urinary 8-oxo-7,8-dihydro-2'-deoxyguanosine (8-oxo-dG). This is a composite outcome studying inflammation and oxidative stress, 2 processes possibly underlying the health effects of air pollutants.
Underlying mechanisms at the molecular level: Mitochondrial DNA damage | Weekly during the 6 week period, changes from baseline measurement are studied
  The mitochondrial DNA content relative to nuclear DNA is determined by qPCR , which is a measure of DNA damage and can give an indication of the need to repair mitochondrial DNA damage.

CONTACTS AND LOCATIONS:
Overall Officials: Tim S Nawrot, PhD, Principal Investigator — Hasselt University
Locations (1):
- Rusthuis Honighsdries, Scherpenheuvel, Limburg, Belgium